CLINICAL TRIAL: NCT02752191
Title: Feraheme As An MRI Contrast Agent For Pediatric Congenital Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paul Finn (Other)
Responsible Party: Sponsor-Investigator, Paul Finn, Professor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-00016
Record Dates: First submitted 2016-04-15; First posted 2016-04-26 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Pediatric Congenital Heart Disease
Keywords: ferumoxytol
MeSH Terms: interventions — Ferrosoferric Oxide; gadofosveset trisodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferumoxytol (Active Comparator): Ferumoxytol, 4mg/kg of body weight, one time infusion of several minutes
  Interventions: Drug: ferumoxytol
- gadofosveset (Active Comparator): gadofosveset, 0.03mmol/kg, one time bolus injection
  Interventions: Drug: gadofosveset

INTERVENTIONS:
Drug: ferumoxytol — ferumoxytol as an MRI contrast agent infused over several minutes
  Other Names: Feraheme
  Arms: Ferumoxytol
Drug: gadofosveset — gadofosveset as an MRI contrast agent injected over several seconds
  Other Names: Ablavar
  Arms: gadofosveset

SUMMARY:
The standard clinical cardiovascular MRI practice for children with CHD frequently involves the use of gadolinium-based contrast agents (GBCA) to enhance tissue contrast. Most GBCAs are small molecules that quickly cross the capillary wall and access the interstitial space, a process which diminishes the signal contrast between blood vessels and surrounding tissue. Therefore, these types of GBCA are most useful for first-pass MR angiography, wherein the images are acquired quickly during the initial 15-30 seconds post-injection when the GBCA concentration is much higher in the arteries than in the interstitial space. For young children with complex CHD, the stringent requirements for high spatial resolution, and the need for cardiac gating and good blood-myocardium contrast in order to provide detailed evaluation of intracardiac structures are not compatible with conventional GBCA-based first-pass MR angiography. Even with Ablavar® (gadofosveset trisodium), an FDA approved GBCA with longer intravascular half-life than other GBCAs, cardiac-gated Ablavar®-enhanced MRI may be insufficient for young children with CHD based on our institutional experience and on data from the literature; there remains diminished blood-tissue contrast during the high-resolution cardiac-gated MRI. Furthermore, there have been safety concerns regarding gadolinium deposition in brain tissues after repeated GBCA exposure as well as concerns of nephrogenic systemic fibrosis (NSF) associated with GBCA injection in young children < 2 years old who may have immature renal function. The long-term health consequences of these effects in the pediatric population are unclear. For the above reasons, we seek to study the diagnostic imaging effectiveness of Feraheme (Feraheme®), an FDA-approved drug for parenteral iron supplementation, as an MRI contrast agent in children with CHD. Although Feraheme® has been approved for the treatment of iron deficiency anemia secondary to renal disease, Feraheme® has been used as an off-label MRI contrast agent at select medical centers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric patients of all ethnicities (age newborn to 6 years) with known or suspected CHD with inconclusive echocardiographic exams and are referred for cardiovascular MRI for further evaluation of cardiac anatomy and function.
* Written informed consent obtained from subject's legal representative/guardian(s) and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Standard clinical contraindications to MRI, including subjects with cochlear implants and implanted cardiac devices
* Subjects with past or current diagnosis of iron overload due to hereditary hemochromatosis or other causes (for subjects receiving Feraheme injection only).
* Subjects with known hypersensitivity or allergy to iron oxide particles.
* Subjects with renal insufficiency defined as estimated glomerular filtration rate (eGFR) < 40 mL/min/1.73m2 (for subjects receiving Ablavar injection only).
* Subjects who are critically ill at the time of MRI and for whom the period of general anesthesia and separation from the critical care nursery or intensive care unit poses added risk as deemed by referring cardiologists, cardiac surgeons or the managing radiologist (for Part II only).
* Other medical conditions, in the judgment of the clinician investigator, that would increase the risks to the child related to participation in the study.

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferumoxytol | Gadofosveset
Started | 14 | 3
Completed | 14 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol | Gadofosveset | Total
Number analyzed (Participants) | 14 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 3 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 6 | 1 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Composite Image Quality Score Among 7 Anatomical Structures.
Description: 1-4 image quality Likert score by an imaging expert, with 4 representing excellent image quality and 1 is non-diagnostic
Time Frame: day 1
Population: Includes all participants that had successfully reconstructed images
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ferumoxytol | Gadofosveset
Number analyzed (Participants) | 13 | 2
score on a scale | 3.9 (0.1) | 2.7 (0.2)

2. Secondary Outcome: Image Quality Score at Individual Anatomical Sites.
Description: 1-4 image quality Likert score by an imaging expert, with 4 representing excellent image quality and 1 is non-diagnostic.
  1. image quality score at the aortic root.
  2. image quality score at the main pulmonary artery.
  3. image quality score at the coronary arteries.
  4. image quality score a the out-flow tracts.
  5. image quality score at the valves.
  6. image quality score at the ventricular chambers.
  7. image quality at the atria.
Time Frame: day 1
Population: includes participants with successfully reconstructed images.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ferumoxytol | Gadofosveset
Number analyzed (Participants) | 13 | 2
score on a scale
  aortic root | 3.8 [3 to 4] | 3 [2 to 4]
  main pulmonary artery | 3.9 [3 to 4] | 3 [3 to 3]
  coronary arteries | 3.8 [3 to 4] | 2.5 [2 to 3]
  outflow tracts | 4 [4 to 4] | 2.5 [2.5 to 2.5]
  valves | 4 [4 to 4] | 2.5 [2.5 to 2.5]
  ventricular chambers | 4 [4 to 4] | 2.8 [2.5 to 3]
  atria | 4 [4 to 4] | 2.8 [2.5 to 3]

3. Secondary Outcome: Incidence of Adverse Events
Description: Number of participants with one or more adverse events
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Gadofosveset
Number analyzed (Participants) | 14 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of MRI exams, typically 1-2 hours
Arm/Group | Ferumoxytol | Gadofosveset
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/3
Other Adverse Events (participants affected / at risk) | 0/14 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT02752191/Prot_SAP_000.pdf